CLINICAL TRIAL: NCT05253508
Title: An Investigation of the Contribution of Proximal Vibratory Cues in Tactile Material Perception'
Brief Title: Propagation Waves in Tactile Material Perception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Collaborators: Delft University of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: NL75084.058.21
Record Dates: First submitted 2022-02-02; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Sensory Processing; Perception; Sense of Touch; Taction
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Repeated-measures design, order randomized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy human participants (Experimental): ring-block anaesthesia with lidocaine in one of the two visits
  Interventions: Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — A digital nerve block by injections to the base of the finger

SUMMARY:
During the exploration of surfaces with the bare finger, vibratory signals arise and propagate through the finger and hand. While research into mechanical and neural response characteristics has demonstrated that these signals carry rich information about touched objects and their properties, only little is known about the role these propagation waves play in human perception and to which extent the somatosensory system is able to collect information from afferents at more proximal locations than the skin-object surface. Using ring-block anaesthesia (lidocaine) we will temporarily inhibit haptic feedback sensations of healthy participants' index finger during interactions with 3D-printed surface probes that are systematically varied in two important material dimensions, namely their roughness and hardness (elasticity), while the participants carry out a well-established psychophysical discrimination task. The results will then be compared to a control condition without anaesthesia. An accelerometer sensor, placed on the dorsal side of the hand, will serve to simultaneously record the propagating tactile waves. Given their role in material perception, thermal cues will be monitored during the experiment with a thermometer and the hydration level of the fingertip skin will be measured regularly using a corneometer. This research will allow us to understand the role of propagation waves in material perception. It seeks to uncover some of the perceptual mechanisms that remain intact during surface discrimination of textured, compliant surfaces, while local information is temporarily inhibited. The results will have implications for how we provide feedback about material properties for sensorimotor control to this living with prosthetic limbs. It is hypothesised that propagation waves that arise during these haptic interactions contain behaviourally relevant information used for the discrimination of surface properties.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* No reported psychiatric or neurological disorders;
* Able to provide informed consent;
* Voluntary participation with written informed consent.

Exclusion Criteria:

* Is pregnant or currently breastfeeding;
* Has a known Lidocaine allergy;
* Is currently undergoing any other medical intervention or taking part in a study involving one;
* Has a history of finger/hand/upper limb trauma or disease;
* Has a disease affecting normal motor functioning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in discrimination thresholds | one year
  The (statistical) difference between psychophysical measures (i.e., difference limen/discrimination thresholds) when the index finger is anaesthetised as compared to non-anaesthetized.

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier Haga Orthopedic Center, Zoetermeer, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided